CLINICAL TRIAL: NCT02674152
Title: A First-in Human Phase I, Non-randomised, Open-label, Multi-center Dose Escalation Trial of BI 836880 Administered by Repeated Intravenous Infusions in Patients With Solid Tumors.
Brief Title: Dose Finding Study of BI 836880 in Patients With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 1336.1; 2014-005395-28 (EudraCT Number)
Record Dates: First submitted 2016-01-04; First posted 2016-02-04 (Estimated); Results first posted 2025-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms

ARMS (5):
- 40 mg BI 836880 (Experimental): BI 836880
  Interventions: Drug: BI 836880
- 120 mg BI 836880 (Experimental): BI 836880
  Interventions: Drug: BI 836880
- 360 mg BI 836880 (Experimental): BI 836880
  Interventions: Drug: BI 836880
- 720 mg BI 836880 (Experimental): BI 836880
  Interventions: Drug: BI 836880
- 1000 mg BI 836880 (Experimental): BI 836880
  Interventions: Drug: BI 836880

INTERVENTIONS:
Drug: BI 836880 — BI 836880

SUMMARY:
This is a Phase I, non-randomized, uncontrolled, open-label, dose escalating study of BI 836880 administered intravenously. The eligible patient population will be patients with advanced solid tumours. At any time during the trial, it will not be permitted to escalate to a dose which does not fulfil the escalation with overdose control (EWOC) criterion

ELIGIBILITY:
Inclusion criteria:

* Age >= 18 years
* Histologically or cytologically confirmed malignancy which is locally advanced or metastatic solid tumor, and either refractory after standard therapy for the disease or for which standard therapy is not reliably effective, e.g. they do not tolerate or have contraindications to otherwise available standard therapy and tumour lesions evaluable for Dynamic contrast-enhanced (DCE)-MRI at MTD.
* ECOG performance status <= 2
* Adequate hepatic, renal and bone marrow functions
* Signed written informed consent.
* Life expectancy min. 3 months in the opinion of the investigator
* Recovery from all reversible adverse events of previous anti-cancer therapies to baseline or CTCAE grade 1, except for alopecia (any grade) sensory peripheral neuropathy CTCAE grade <= 2 or considered not clinically significant.
* adequate contraception by male and female patient during the trial and for at least 6 months after end of treatment.

Exclusion criteria:

* Known hypersensitivity to the trial drugs or their excipients
* Current or prior treatment with any systemic anti-cancer therapy either within 28 days or a minimum of 5 half-lives, whichever is shorter of trial onset.
* Serious concomitant disease, especially those affecting compliance with trial requirements or which are considered relevant for the evaluation of the endpoints of the trial drug
* Major injuries and/or surgery or bone fracture within 4 weeks of start of treatment, or planned surgical procedures during the trial period.
* patients with personal or family history of QT prolongation and/or long QT syndrome, or prolonged QTcF at baseline (> 470 ms). QTcF will be calculated by Investigator as the mean of the 3 ECGs taken at screening.
* Significant cardiovascular/cerebrovascular diseases (i.e. uncontrolled hypertension, unstable angina, history of infarction within past 6 months, congestive heart failure > NYHA II). Uncontrolled hypertension defined as: blood pressure in rested and relaxed condition >=140 mmHg systolic, or >=90 mmHg diastolic (with or without medication), measured according to protocol.
* History of severe haemorrhagic or thromboembolic event in the past 12 months (excluding central venous catheter thrombosis and peripheral deep vein thrombosis).
* Known inherited predisposition to bleeding or to thrombosis in the opinion of the investigator.
* Patient with brain metastases that are symptomatic and/or require therapy.
* Patients who require full-dose anticoagulation (according to local guidelines).
* Active alcohol or drug abuse in the opinion of the investigator.
* Patients who are under judicial protection and patients who are legally institutionalized.
* Patients unable or unwilling to comply with protocol
* Women who are pregnant, nursing, or who plan to become pregnant while in the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2016-01-05 (Actual); Primary Completion 2018-09-12 (Actual); Study Completion 2020-11-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (3):
- INS Curie, Paris, France
- Germany (2):
  - Universitätsklinikum Augsburg, Augsburg
  - Universitätsklinikum Freiburg, Freiburg im Breisgau

REFERENCES:
- [Derived] Keller S, Kunz U, Schmid U, Beusmans J, Buchert M, He M, Jayadeva G, Le Tourneau C, Luedtke D, Niessen HG, Oum'hamed Z, Pleiner S, Wang X, Graeser R. Comprehensive biomarker and modeling approach to support dose finding for BI 836880, a VEGF/Ang-2 inhibitor. J Transl Med. 2024 Oct 14;22(1):934. doi: 10.1186/s12967-024-05612-x. PMID 39402675
- [Derived] Le Tourneau C, Becker H, Claus R, Elez E, Ricci F, Fritsch R, Silber Y, Hennequin A, Tabernero J, Jayadeva G, Luedtke D, He M, Isambert N. Two phase I studies of BI 836880, a vascular endothelial growth factor/angiopoietin-2 inhibitor, administered once every 3 weeks or once weekly in patients with advanced solid tumors. ESMO Open. 2022 Oct;7(5):100576. doi: 10.1016/j.esmoop.2022.100576. Epub 2022 Sep 13. PMID 36108560
- See also: Related Info — https://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A non-randomized, open-label, multi-center dose escalation trial to determine the maximum tolerated dose and recommended Phase 2 dose of BI 836880 in patients with advanced or metastatic/refractory solid tumours.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria.
  Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Groups:
- 40 mg BI 836880: 40 milligrams (mg) BI 836880 solution for infusion were administered intravenous as rate-controlled infusion once per treatment cycle (21 days) in patients with advanced or metastatic solid tumour. Administration was continued until disease progression or until intolerable toxicities had been observed, up to 786 days. The pharmaceutical formulation was diluted with 50ml/vial to prepare solution for infusion of BI 836880.
- 120 mg BI 836880: 120 mg BI 836880 solution for infusion were administered intravenous as rate-controlled infusion once per treatment cycle (21 days) in patients with advanced or metastatic solid tumour. Administration was continued until disease progression or until intolerable toxicities had been observed, up to 786 days. The pharmaceutical formulation was diluted with 50ml/vial to prepare solution for infusion of BI 836880.
- 360 mg BI 836880: 360 mg BI 836880 solution for infusion were administered intravenous as rate-controlled infusion once per treatment cycle (21 days) in patients with advanced or metastatic solid tumour. Administration was continued until disease progression or until intolerable toxicities had been observed, up to 786 days. The pharmaceutical formulation was diluted with 50ml/vial to prepare solution for infusion of BI 836880.
- 720 mg BI 836880: 720 mg BI 836880 solution for infusion were administered intravenous as rate-controlled infusion once per treatment cycle (21 days) in patients with advanced or metastatic solid tumour. Administration was continued until disease progression or until intolerable toxicities had been observed, up to 786 days. The pharmaceutical formulation was diluted with 50ml/vial to prepare solution for infusion of BI 836880.
- 1000 mg BI 836880: 1000 mg BI 836880 solution for infusion were administered intravenous as as rate-controlled infusion once per treatment cycle (21 days) in patients with advanced or metastatic solid tumour. Administration was continued until disease progression or until intolerable toxicities had been observed, up to 786 days. The pharmaceutical formulation was diluted with 50ml/vial to prepare solution for infusion of BI 836880.
Period: Overall Study
Arm/Group | 40 mg BI 836880 | 120 mg BI 836880 | 360 mg BI 836880 | 720 mg BI 836880 | 1000 mg BI 836880
Started (Treated) | 3 | 2 | 2 | 17 | 5
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 2 | 2 | 17 | 5
Not completed — Personal Reasons | 1 | 0 | 0 | 1 | 1
Not completed — Other adverse event or clinical progression | 0 | 1 | 0 | 3 | 0
Not completed — Dose-limiting toxicity | 0 | 0 | 0 | 0 | 1
Not completed — Progressive Disease | 2 | 1 | 1 | 13 | 2
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Treated Set (TS): The TS included all patients enrolled in the trial who were documented to have taken at least 1 dose of trial medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | 40 mg BI 836880 | 120 mg BI 836880 | 360 mg BI 836880 | 720 mg BI 836880 | 1000 mg BI 836880 | Total
Number analyzed (Participants) | 3 | 2 | 2 | 17 | 5 | 29
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.7 (8.1) | 70.5 (6.4) | 47.0 (9.9) | 56.7 (14.2) | 49.4 (13.2) | 55.8 (13.4)
Sex: Female, Male [Count of Participants; unit: Participants] — Treated Set (TS): The TS included all patients enrolled in the trial who were documented to have taken at least 1 dose of trial medication.
  Participants
    Female | 1 | 1 | 1 | 12 | 3 | 18
    Male | 2 | 1 | 1 | 5 | 2 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 1 | 1 | 3 | 3 | 9
  Unknown or Not Reported | 2 | 1 | 1 | 14 | 2 | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 1 | 1 | 1 | 3 | 3 | 9
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 1 | 14 | 2 | 20

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD)
Description: Maximum tolerated dose (MTD) defined as the highest dose with less than 25% risk of the true dose-limiting toxicity (DLT) rate being above 0.33 during the MTD evaluation period, defined as 3 weeks after first administration of trial medication (i.e. cycle 1). Patients who did not complete the MTD evaluation period for reasons other than DLT were excluded from the analysis of the primary endpoint.
Time Frame: Up to 3 weeks after the first administration of trial medication.
Population: Dose-finding cohort treated set: All patients enrolled in dose finding and confirmation of MTD cohort of the trial who were documented to have taken at least 1 dose of study medication and were evaluable for the MTD determination.
Measure: Number; unit: Milligram
Groups:
- BI 836880 - All Dose Groups: 40/120/360/720 or 1000 mg BI 836880 solution for infusion were administered intravenous as rate-controlled infusion once per treatment cycle (21 days) in patients with advanced or metastatic solid tumour. The pharmaceutical formulation was diluted with 50ml/vial to prepare solution for infusion of BI 836880.
Arm/Group | BI 836880 - All Dose Groups
Number analyzed (Participants) | 17
Milligram | 720

2. Primary Outcome: Number of Patients With Dose-limiting Toxicities (DLT) in the Maximum Tolerated Dose (MTD) Period
Description: DTLs are defined as followed:
  * Drug-related Common Terminology Criteria for Adverse Events (CTCAE) grade ≥3 non-haematological toxicity
  * CTCAE Grade 4 neutropenia lasting >7 days or complicated by infection (please note that in case of grade 4 neutropenia a more frequent follow up of patient was necessary
  * Febrile neutropenia of CTCAE Grade ≥3
  * CTCAE Grade 4 thrombocytopenia or CTCAE Grade ≥3 thrombocytopenia with bleeding
  * Treatment delay for >2 weeks due to unresolved drug-related AEs, which started within 3 weeks after the first treatment
  * Hypertension: increase of diastolic blood pressure (DBP) by 15 millimetre of mercury (mmHg) confirmed by a second measurement or by ambulatory blood pressure measurement (when indicated, e.g. white coat effect) which could not be controlled by hypertensive medication and required a dose reduction of BI 836880 for further treatment cycle
  * Proteinuria: urinary protein ≥3.5 gram/day (CTCAE Grade 3)
Time Frame: Up to 3 weeks after the first administration of trial medication.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 40 mg BI 836880 | 120 mg BI 836880 | 360 mg BI 836880 | 720 mg BI 836880 | 1000 mg BI 836880
Number analyzed (Participants) | 2 | 2 | 2 | 7 | 4
Participants | 0 | 0 | 0 | 0 | 1

3. Secondary Outcome: Number of Patients With Drug-related Adverse Events Leading to Dose Reduction or Discontinuation During Treatment Period
Description: Number of patients with drug-related adverse events leading to dose reduction or discontinuation during treatment period.
Time Frame: From first drug infusion until 42 days (residual effect period) after last drug infusion, up to 828 days.
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | 40 mg BI 836880 | 120 mg BI 836880 | 360 mg BI 836880 | 720 mg BI 836880 | 1000 mg BI 836880
Number analyzed (Participants) | 3 | 2 | 2 | 17 | 5
Participants | 0 | 0 | 0 | 1 | 1

4. Secondary Outcome: Area Under the Serum Concentration-time Curve Over the Time Interval From 0 Extrapolated to Infinity (AUC0-tz) After the First Dose
Description: Area under the serum concentration-time curve over the time interval from 0 extrapolated to infinity (AUC0-tz) after the first dose.
Time Frame: 5 minutes before start of BI 836880 infusion and immediately after end of infusion (i.e. 1.5 hours (h) after start of infusion) and 2h, 3h, 5h, 8h, 24h, 72h, 168h, 336h and 504h after start of BI 826880 infusion in cycle 1.
Population: Pharmacokinetic (PK) analysis set: All patients who were treated and provided at least 1 observation for at least 1 PK endpoint without an important protocol deviation relevant to PK evaluations.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram * hours/ milliliter
Arm/Group | 40 mg BI 836880 | 120 mg BI 836880 | 360 mg BI 836880 | 720 mg BI 836880 | 1000 mg BI 836880
Number analyzed (Participants) | 3 | 2 | 2 | 17 | 5
Microgram * hours/ milliliter | 2180 (152) | 4100 (38.7) | 15000 (71.1) | 32900 (28.1) | 40000 (66.6)

5. Secondary Outcome: Terminal Half-life (t_1/2) of BI 836880
Description: Terminal half-life (t_1/2) of BI 836880.
Time Frame: as for outcome 4
Population: Pharmacokinetic (PK) analysis set: All patients who were treated and provided at least 1 observation for at least 1 PK endpoint without an important protocol deviation relevant to PK evaluations. Only participants with available data were included in the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | 40 mg BI 836880 | 120 mg BI 836880 | 360 mg BI 836880 | 720 mg BI 836880 | 1000 mg BI 836880
Number analyzed (Participants) | 2 | 2 | 2 | 16 | 4
Hours | 241 (16.3) | 210 (5.07) | 265 (7.42) | 289 (19.1) | 279 (8.96)

ADVERSE EVENTS:
Time Frame: From first drug infusion until 42 days (residual effect period) after last drug infusion, up to 828 days. For all-cause mortality: From signing informed consent, until end of trial, up to 1546 days.
Description: Treated Set (TS): The TS included all patients enrolled in the trial who were documented to have taken at least 1 dose of study medication.
Groups:
- Total BI 836880: 40/120/360/720 or 1000 mg BI 836880 solution for infusion were administered intravenous as rate-controlled infusion once per treatment cycle (21 days) in patients with advanced or metastatic solid tumour. The pharmaceutical formulation was diluted with 50ml/vial to prepare solution for infusion of BI 836880.
Arm/Group | 40 mg BI 836880 | 120 mg BI 836880 | 360 mg BI 836880 | 720 mg BI 836880 | 1000 mg BI 836880 | Total BI 836880
All-Cause Mortality (participants affected / at risk) | 2/3 | 1/2 | 0/2 | 4/17 | 2/5 | 9/29
Serious Adverse Events (participants affected / at risk) | 1/3 | 2/2 | 1/2 | 6/17 | 5/5 | 15/29
Other Adverse Events (participants affected / at risk) | 3/3 | 2/2 | 2/2 | 17/17 | 5/5 | 29/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 40 mg BI 836880 (N=3) | 120 mg BI 836880 (N=2) | 360 mg BI 836880 (N=2) | 720 mg BI 836880 (N=17) | 1000 mg BI 836880 (N=5) | Total BI 836880 (N=29)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 1
Myocarditis (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 2
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Mechanical ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Subileus (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Death (General disorders) | 0 | 1 | 0 | 0 | 0 | 1
Impaired healing (General disorders) | 0 | 0 | 0 | 0 | 1 | 1
Pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 1
Bile duct stone (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 1
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 1
Hepatic pain (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 1
Hepatomegaly (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 1
Device related infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 2
Peritonitis bacterial (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 1
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 40 mg BI 836880 (N=3) | 120 mg BI 836880 (N=2) | 360 mg BI 836880 (N=2) | 720 mg BI 836880 (N=17) | 1000 mg BI 836880 (N=5) | Total BI 836880 (N=29)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 6 | 2 | 8
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 1
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 2 | 1 | 4
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2 | 0 | 2
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1 | 1 | 0 | 2
Hypothyroidism (Endocrine disorders) | 0 | 0 | 1 | 0 | 2 | 3
Dry eye (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 1
Eyelid haematoma (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 0 | 3 | 2 | 7
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 2 | 1 | 4
Aphthous ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Constipation (Gastrointestinal disorders) | 1 | 0 | 1 | 5 | 1 | 8
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 1 | 5 | 1 | 8
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Enterocutaneous fistula (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 2
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 1 | 3
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Melaena (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 9 | 3 | 13
Odynophagia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Oesophageal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1 | 1 | 6 | 2 | 11
Asthenia (General disorders) | 2 | 0 | 1 | 10 | 2 | 15
Chest pain (General disorders) | 0 | 0 | 0 | 1 | 2 | 3
Chills (General disorders) | 0 | 0 | 0 | 1 | 0 | 1
Face oedema (General disorders) | 1 | 0 | 1 | 0 | 0 | 2
Fatigue (General disorders) | 0 | 0 | 1 | 0 | 0 | 1
Hernia (General disorders) | 0 | 0 | 0 | 0 | 1 | 1
Impaired healing (General disorders) | 0 | 0 | 0 | 0 | 1 | 1
Localised oedema (General disorders) | 0 | 1 | 0 | 0 | 0 | 1
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 1 | 0 | 1
Oedema peripheral (General disorders) | 0 | 0 | 1 | 4 | 2 | 7
Pain (General disorders) | 0 | 1 | 0 | 1 | 0 | 2
Peripheral swelling (General disorders) | 0 | 0 | 0 | 0 | 1 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 3 | 0 | 3
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 1
Hepatic pain (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 1
Hepatotoxicity (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 1
Allergy to immunoglobulin therapy (Immune system disorders) | 0 | 0 | 0 | 1 | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 3 | 0 | 3
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 2
Influenza (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1 | 1 | 2 | 4
Oral fungal infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 2
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Urinary tract infection (Infections and infestations) | 0 | 1 | 1 | 2 | 2 | 6
Bone contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1 | 2
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 4 | 1 | 5
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 1
Stoma site inflammation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 1
Stoma site rash (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 1
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 1
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 0 | 0 | 1 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 2 | 3 | 5
Amylase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 7 | 2 | 9
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 1 | 2 | 3
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 3 | 2 | 5
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 1 | 1 | 2
C-reactive protein increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1
Electrocardiogram T wave inversion (Investigations) | 0 | 0 | 1 | 0 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1
Lipase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1
Weight decreased (Investigations) | 0 | 0 | 1 | 0 | 1 | 2
Acidosis (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 2
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 1
Iron deficiency (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 3 | 2 | 6
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 1 | 1 | 4
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1
Trismus (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 1 | 2
Dysaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 1
Depression (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 1 | 0 | 2
Mixed anxiety and depressive disorder (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 1
Haematuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 1
Micturition urgency (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 1 | 1 | 1 | 0 | 3
Renal failure (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 1
Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 1
Female genital tract fistula (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 1 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 4 | 0 | 6
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0 | 2
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 2
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 0 | 2
Hypertension (Vascular disorders) | 3 | 2 | 2 | 15 | 4 | 26
Lymphoedema (Vascular disorders) | 0 | 0 | 0 | 1 | 1 | 2
Raynaud's phenomenon (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2019-03-08): https://cdn.clinicaltrials.gov/large-docs/52/NCT02674152/Prot_000.pdf
  • Statistical Analysis Plan (2017-06-21): https://cdn.clinicaltrials.gov/large-docs/52/NCT02674152/SAP_001.pdf